CLINICAL TRIAL: NCT05421546
Title: Characterisation of the Effects of Spermidine, a Nutrition Supplement, on the Immune Memory Response to Coronavirus Vaccine in Older People
Brief Title: Improving Vaccination in Older Adults by Inducing Autophagy With Spermidine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: R75468/RE001
Record Dates: First submitted 2022-06-13; First posted 2022-06-16 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2022-08

CONDITIONS: COVID-19; Vaccine Reaction
MeSH Terms: conditions — COVID-19 | interventions — Spermidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spermidine arm (Active Comparator): This arm will enrol 20 volunteers aged 65 years of age or older (65-90) who have received two doses of the Coronavirus vaccine, with the vaccination course completed more than 8 weeks before recruitment. Following a baseline venous blood sample, participants will receive Spermidine supplements 6mg/day and oral administration once daily. A research appointment and venous blood sample will be requested at the point of recruitment, 5 weeks, 13 weeks and 37 weeks after recruitment of the participant.
  Interventions: Dietary Supplement: Spermidine or Placebo
- Placebo arm (Placebo Comparator): This arm will enrol 20 volunteers aged 65 years of age or older (65-90) who have received two doses of the Coronavirus vaccine, with the vaccination course completed more than 8 weeks before recruitment. Following a baseline venous blood sample, participants will receive placebo oral administration once daily. A research appointment and venous blood sample will be requested at the point of recruitment, 5 weeks, 13 weeks and 37 weeks after recruitment of the participant.
  Interventions: Dietary Supplement: Spermidine or Placebo

INTERVENTIONS:
Dietary Supplement: Spermidine or Placebo — The supplement, Spermidine, is made mainly from wheatgerm and can be bought in health food shops. It is a powder that can be easily dissolved in water and taken as a drink. The 'placebo' is a sugar powder that can be similarly dissolved in water and taken as a drink.

SUMMARY:
Easing the morbidity and economic burden of age-related diseases is one of the major medical challenges. One of the key obstacles to healthy ageing is immune senescence, including the failure of lymphocytes to respond adequately to infection, malignancy and vaccination. Infectious diseases remain the fourth most common cause of death among the elderly in the developed world. Moreover, the gain of chronic low-grade non-specific inflammation with age contributes to many age-related diseases. Our early work showed that autophagy, the main cellular bulk degradation pathway in the cell, prevents ageing of the immune system. In preclinical models we showed an age-related decline in T cell autophagy. We rejuvenated the immune system by restoring autophagy in T and B cells with the autophagy-inducing metabolite spermidine. Here we are asking for matched funds for a small human clinical trial to confirm that spermidine has the same effect when administered to humans. We will give the nutraceutical spermidine to human volunteers aged >65 years either during or after vaccination against SARS-CoV-2 or influenza to test improvement of vaccine responses, immune senescence and inflamm-aging. We will also confirm whether a novel pathway we discovered that links spermidine to autophagy operates in humans, allowing us to make more specific drugs in the future. This small study of 120 volunteers overall will pave the way for a larger clinical trial with spermidine or novel related drugs.

DETAILED DESCRIPTION:
The outbreak of SARS-CoV-2 and coronavirus disease (COVID-19) has caused a great threat to global public health with the majority of deaths occurring in older adults. The development of effective treatments and vaccines against COVID-19 has become a pressing and urgent challenge to overcome. Successful protective immune responses stimulated by vaccination of older people (people aged greater than 65 years old) against pathogens is considered one of the big challenges in our society.

Immune senescence is thought to be important in the reduced immune response that has been widely observed, following immunization of older adults. This is characterized by poor induction and recall of B and T cell memory responses upon exposure to viruses and vaccines.

Most vaccines are less immunogenic effective in the older population, in particular influenza vaccines. Autophagy is thought to be one of the few cellular processes that underlie many facets of cellular aging including immune senescence. Autophagy delivers 'unwanted' cytoplasmic material to lysosomes inside a cell for degradation. Autophagy also limits mitochondrial dysfunction and accumulation of reactive oxygen species (ROS).

Deletion of key autophagy genes leads to a change in cellular immunity, with loss of function in mouse memory CD8+ T cells, hematopoietic stem cells, and macrophages. We have seen that autophagy levels also decline with age in human peripheral CD8+ T cells and correlate with vaccine responses.

Importantly, we have demonstrated that we can improve CD8+ T memory responses in aged mice with a supplement called spermidine. Spermidine is a metabolite synthesised from arginine. It is commonly found in wheatgerm and soya and is available in the United Kingdom (UK) as a nutritional food supplement, often described as a polyamine. It's safety and tolerability has been studied and no adverse effects have been demonstrated and it is readily available to buy from mainstream retail companies e.g. Amazon. Our data showed for the first time that autophagy is indeed highly active in human CD8+ T cells in two different experimental vaccination trials. Polyamine levels also fall with age in peripheral mononuclear cells. When supplemented with spermidine, the autophagic function can be rejuvenated in CD8+ T cells from old donors, and levels of the important effector molecules increased. As a consequence, the immune response is enhanced.

Moreover, autophagy and effector function are maintained by spermidine in T cells from young donors. This demonstrates that the function of human CD8+ T cells can be improved with spermidine. Taken together with our previous work on B cells, this leads us to the hypothesis that both T and B cell responses to infections and vaccinations are exquisitely reliant on sufficient autophagy levels, which are maintained by intracellular spermidine. This work highlights the potential of spermidine as a vaccine adjuvant in the older adults.

This phase 1, double-blinded, randomised controlled trial is designed as a feasibility study to examine the safety of Spermidine supplements and its effects on the immune response (antibodies) to COVID vaccine in older people.

AIMS AND OBJECTIVES The primary objective of this feasibility study is to determine the safety of daily Spermidine supplements following vaccination for Coronavirus (SARS-CoV-2) and a booster and its effects on antibody levels in older people, using validated assays.

Our secondary objective is to determine the effects of daily Spermidine supplements on the immune 'memory' response to Coronavirus vaccine and a booster in older people. We will examine if Spermidine improves the duration of the antibody-mediated immune response after the Coronavirus vaccine/booster with validated assays and then determine the molecular and immunological signature driving immunity. We will also use data collected to perform a power calculation for future larger studies.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 65 years old or more and must have the capacity to provide written consent after discussing the participant information sheet with a member of the clinical study team. Participants must have received 2 doses of the COVID vaccine and a booster dose.

Exclusion Criteria:

* Participants who are acutely unwell.
* Participants who have had a clear clinical history of COVID symptoms or a previous positive COVID PCR( polymerase chain reaction) swab or antibody test
* Participants who cannot provide informed written consent
* Participants who use systemic steroids for more than one week e.g prednisolone >0.5mg/kg/day in the three months prior to first study intervention
* Chronic administration (≥14 days in total) of immunosuppressants or other immune modifying drugs in the 3 months prior to first study intervention
* Receipt of blood, blood products and/or plasma derivatives or any immunoglobulin preparation in the three months prior to first study intervention
* Participants who have been diagnosed with medical conditions that can suppress the immune system or diabetes
* Participants with previous allergy to or constituent parts of Spermidine supplements or who have gluten intolerance
* Participants already taking Spermidine supplements at the time of recruitment or for 6 months prior to recruitment to the study
* Participants that are in custody
* Participants that do not live in the UK
* Participants that are pregnant
* Participants who are shielding

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-12-02 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to determine the safety of daily Spermidine supplements following the vaccine booster for Coronavirus (SARS-CoV-2) and its effects on antibody levels in older people, using validated assays. | 37 weeks
  1. The safety of daily Spermidine supplements following the vaccine booster for Coronavirus (SARS-CoV-2).
  2. The SARS-CoV-2 antibody levels in older people, using validated assays.

SECONDARY OUTCOMES:
Our secondary objective is to determine the effects of daily Spermidine supplements on the immune 'memory' response to Coronavirus vaccine and the booster in older people. | 37 weeks
  1. Longevity of immune 'memory' response to SARS-CoV-2 vaccine measuring antibody and T cell responses.

CONTACTS AND LOCATIONS:
Overall Officials: Katja Simon, Prof., Principal Investigator — University of Oxford
Locations (1):
- University of Oxford, Oxford, United Kingdom